CLINICAL TRIAL: NCT03251716
Title: Berberine in the Treatment of Metabolic Syndrome : an Open Label Clinical Study in Female Schizophrenia Patients
Brief Title: Berberine Treat Metabolic Syndrome in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ber-open-2015-TJAH
Record Dates: First submitted 2017-08-03; First posted 2017-08-16 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2017-12

CONDITIONS: Metabolic Syndrome; Female; Schizophrenia
Keywords: Metabolic syndrome; Schizophrenia; Efficacy; Female; Berberine
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia | interventions — Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- berberine adjunctive group (Experimental): Only one treatment group in this study, without a preset control group,subjects who meet the criteria will entere the berberine adjunctive group
  Interventions: Drug: berberine

INTERVENTIONS:
Drug: berberine — berberine 300mg TID add-on for berberine adjunctive group
  Other Names: berberine hydrochloride

SUMMARY:
In early clinical study investigators confirmed that berberine could prevent glucose and lipid metabolism disorder in schizophrenia, so investigators intend to verify the effect and safety of berberine in treatment for metabolic syndrome in schizophrenia.

DETAILED DESCRIPTION:
This study is an open lable clinical intervention trial, include 30 female subjects with diagnosis of schizophrenia and metabolic syndrome.Participants will be given berberine（ 300mgTID） as an add-on therapy lasting 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. subjects with the diagnosis of schizophrenia depend on Statistical Manual, Fifth Edition (DSM-5) ;
2. Female subjects aged 18-60 years;
3. monotherapy of atypical antipsychotics for 2 weeks or more , including olanzapine, clozapine, risperidone, and perphenazine；
4. subjects with diagnosis of metabolic syndrome depending on guidelines for the prevention and treatment of dyslipidemia in Chinese adults in 2007;
5. the subjects and their guardians sign the informed consent agreement.

Exclusion Criteria:

1. subjects with diagnosis of other psychiatric disorders except schizophrenia depend on DSM-5;
2. chronic organic diseases involving any central nervous system, such as tumors and inflammation, brain trauma, active seizures, vascular diseases, Parkinson's disease, myasthenia gravis, and other degenerative diseases;
3. a history of gastrointestinal surgery or the presence of any possibility of interfering with the absorption, distribution, metabolism, or excretion of drugs situation;
4. used long-acting antipsychotic drugs or receive electroconvulsive therapy (MECT) or receive transcranial magnetic stimulation therapy in the last 1 months;
5. serious physical diseases, including uncontrolled hypertension, severe cardiovascular, cerebrovascular, and pulmonary diseases, thyroid diseases, etc;
6. currently receiving anti-inflammatory or immunosuppressive treatment, including oral steroids;
7. a history of chronic infection, including tuberculosis, AIDS and hepatitis;
8. allergic to berberine,or hemolytic anemia or glucose -6- phosphate dehydrogenase deficiency;
9. pregnant women, lactating women；
10. participants were involved in other clinical trials within 1 months prior to the signing of informed consent
11. other reasons judged by the researchers to be inappropriate for the clinical study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change of FBG | Change from Baseline serum fasting biood glucose at 8 weeks
  Serum fasting biood glucose

SECONDARY OUTCOMES:
Change of TG | Change from Baseline serum triglyceride at 8 weeks
  Serum triglyceride
Change of LDL | Change from Baseline serum low density lipoprotein at 8 weeks
  Serum low density lipoprotein
Change of BP | Change from Baseline Systolic Blood Pressure at 8 weeks
  Systolic blood pressure
Change of waist | Change from Baseline waistline at 8 weeks
  Waistline
Change of BP | Change from Baseline Diastolic Blood Pressure at 8 weeks
  Diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China